CLINICAL TRIAL: NCT01538199
Title: Evaluation of LED Therapeutic Effect in Depression (ELATED): a Placebo-Controlled, Parallel Study of Efficacy, Tolerability and Acceptability of a Novel Approach in the Community
Brief Title: Transcranial Laser Therapy for Major Depressive Disorder
Acronym: ELATED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paolo Cassano (Other)
Collaborators: Mclean Hospital (Other); North Suffolk Mental Health Association (Other)
Responsible Party: Sponsor-Investigator, Paolo Cassano, Staff Psychiatrist, Depression Clinical & Research Program (DCRP), Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010P002718; 2010A050442 (Other: Harvard Medical School)
Record Dates: First submitted 2012-02-17; First posted 2012-02-24 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-10

CONDITIONS: Major Depressive Disorder
Keywords: Device study; Depression; Major Depression; Major Depressive Disorder; MDD; Device for depression; Alternatives to medication for depression; Massachusetts General Hospital; Boston
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TLT Treatment Group 1 (Experimental): The TLT group will receive 2 near-infrared radiation via Transcranial LED Therapy (TLT) treatments per week for 8 weeks
  Interventions: Device: Near-infrared radiation via Transcranial LED Therapy
- TLT Treatment Group 2 (Sham Comparator): The sham group will receive 2 treatments of the sham device per week for 8 weeks
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Near-infrared radiation via Transcranial LED Therapy — The subject will lie down comfortably on a exam bed . The sites of application of TLT (left and right forehead) will be inspected for any skin lesions (e.g. laceration or signs of inflammation) which would contraindicate the treatment. The subject will wear protective eyewear in the form of goggles or eye pads.
  The staff administering the TLT will be careful not to shine the light in or near the eyes of the subject. The two OLS devices will be secured in position with the use of a Hair Net. The delivery of the TLT is expected to last 20 min total (simultaneous application on the left and right forehead). The subject will be asked to rest for five minutes after the delivery of TLT. The skin at the sites of the application will be inspected again prior to dismissing the subject.
  Other Names: PhotoMedex Omnilux New-U; Near-infrared radiation (NIR)
  Arms: TLT Treatment Group 1
Device: Sham device — The sham device does not emit near-infrared radiation.
  Other Names: PhotoMedex Omnilux New-U.
  Arms: TLT Treatment Group 2

SUMMARY:
The purpose of this study is to see if using Transcranial LED Therapy (TLT) using the PhotoMedex's Omnilux NEw-U LED helps improve symptoms of major depressive disorder (MDD). TLT works by briefly delivering near-infrared (non-visible) radiations to the forehead. The radiations penetrate the brain and stimulate the cells & metabolism.

Our goals are

* To assess the antidepressant effect of the TLT in depressed subjects.
* To assess the safety and tolerability of the TLT in depressed subjects
* To assess the acceptability of the TLT in depressed subjects
* To pilot test the impact on cognition of the TLT in depressed subjects (Ancillary Study)

DETAILED DESCRIPTION:
TLT has previously been evaluated in two large studies of people who have had a stroke. To date, TLT has been administered to over 550 people who have had a stroke. TLT has also been used in 10 people with MDD who were taking part in a research study. During this study, TLT was shown to relieve MDD symptoms without causing too many side effects.

The -Infrared Radiation (NIR) device is also marketed for wrinkles treatment, however it is experimental for the use in depression. An experimental device means that it is one that has not been approved by the U.S. Food and Drug Administration (FDA).

During this study, the investigators hope to better find out if NIR TLT is helpful for treating depression. The investigators will do this by comparing the effects of TLT ("active treatment") NIR device to a sham treatment (which is an inactive or "pretend" treatment) device. The sham ("pretend") device looks exactly like the NIR device but will not use a near-infrared radiation during the study visits. There are two sets of identical devices that will be used in this study, producing active and sham treatment, respectively. The devices work exactly the same when you are receiving active treatment and sham treatment, except that the devices will produce therapeutic transcranial LED energy during the active treatment sessions but it will not produce this LED energy during the sham treatment sessions.

The investigators hope to enroll about 30 subjects in this study at the Massachusetts General Hospital Depression Clinical and Research Program.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 18 years of age at screening, but has not had their 66th birthday.
* SCID diagnosis of major depressive disorder (Structured Clinical Interview for Diagnostic Statistical Manual-IV)
* HAM-D-17 >14 and < 25
* Women of child-bearing potential must use a double-barrier method for birth control (e.g. condoms with spermicide) if sexually active.
* Subject Informed Consent obtained in writing in compliance with local regulations prior to enrollment into this study.
* The subject (and caregiver, if applicable) is willing to participate in this study for at least 8 weeks.
* Subjects on an antidepressant will need to be on a stable dose for at least six weeks.

Exclusion Criteria:

* The subject is pregnant or lactating.
* The subject failed two or more FDA-approved antidepressants during current episode
* Subjects with less than 2 months MDD symptom free prior to current episode.
* The subject used targeted psychotherapies for depression during current episode (support therapy or counseling are allowed)
* Substance dependence or abuse in the past 6 months
* Psychotic disorder or psychotic episode (current psychotic episode per SCID assessment)
* Bipolar affective disorder (per SCID assessment)
* Unstable medical illness, defined as any medical illness which has not been well-controlled with standard-of-care medications (e.g., insulin for diabetes mellitus, HCTZ for hypertension)
* Active suicidal or homicidal ideation, as determined by CHRT screening
* The subject has a significant skin condition (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo) on the subject's scalp that is found to be directly below any of the procedure sites.
* The subject has an implant of any kind in the head (e.g. stent, clipped aneurysm, embolised AVM, implantable shunt - Hakim valve).
* Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment (in US: Visudine (verteporfin) - for age related macular degeneration; Aminolevulinic Acid- for actinic keratoses; Photofrin (porfimer sodium) - for esophageal cancer, non-small cell lung cancer; Levulan Kerastick (aminolevulinic acid HCl) - for actinic keratosis; 5-aminolevulinic acid (ALA)- for non-melanoma skin cancer)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Cassano, MD, PhD, Principal Investigator — Massachusetts General Hospital, Harvard Medical School, and North Suffolk Mental Health Association
Locations (2):
- United States (2):
  - Massachusetts General Hospital- Depression Clinical and Research Program, Boston, Massachusetts
  - Chelsea Counseling Center- North Suffolk Mental Health Association, Chelsea, Massachusetts

REFERENCES:
- [Derived] Cassano P, Cusin C, Mischoulon D, Hamblin MR, De Taboada L, Pisoni A, Chang T, Yeung A, Ionescu DF, Petrie SR, Nierenberg AA, Fava M, Iosifescu DV. Near-Infrared Transcranial Radiation for Major Depressive Disorder: Proof of Concept Study. Psychiatry J. 2015;2015:352979. doi: 10.1155/2015/352979. Epub 2015 Aug 19. PMID 26356811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in 2012 for the pilot phase of the study. Participants were recruited from February 2014 through June 2015 via Craigslist advertisements and the general research phone line for the Depression Clinical and Research Program at Massachusetts General Hospital.
Pre-assignment Details: 10 subjects from the pilot phase and 9 subjects from phase 2 screen failed (HAM-D scores below or above threshold, active substance abuse, exclusionary comorbid medical disorder, did not pass drug screen, just started psychotherapy). 6 participants dropped out after screen (time constraints, moving, LTFU). 1 subject had primary diagnosis of PTSD.
Groups:
- TLT Treatment Group 1 (Active TLT Treatment): The TLT group will receive 2 near-infrared radiation via Transcranial LED Therapy (TLT) treatments per week for 8 weeks
  Near-infrared radiation via Transcranial LED Therapy: The subject will lie down comfortably on a exam bed . The sites of application of TLT (left and right forehead) will be inspected for any skin lesions (e.g. laceration or signs of inflammation) which would contraindicate the treatment. The subject will wear protective eyewear in the form of goggles or eye pads.
  The staff administering the TLT will be careful not to shine the light in or near the eyes of the subject. The two OLS devices will be secured in position with the use of a Hair Net. The delivery of the TLT is expected to last 20 min total (simultaneous application on the left and right forehead). The subject will be asked to rest for five minutes after the delivery of TLT. The skin at the sites of the application will be inspected again prior to dismissing the subject.
- TLT Treatment Group 2 (Placebo): The sham group will receive 2 treatments of the sham device per week for 8 weeks
  Sham device: The sham device does not emit near-infrared radiation.
- Pilot Study Treatment Group 1: The TLT group will receive 2 TLT treatments per week for 3 weeks followed by a cross-over phase (where no treatment is given), followed by 2 sham treatments per week for 3 weeks.
  (see protocol change 10/28/2014)
- Pilot Study Treatment Group 2: The sham group will receive 2 sham treatments per week for 3 weeks followed by a cross-over phase (where no treatment is given), followed by 2 TLT treatments per week for 3 weeks.
  (see protocol change 10/28/2014)
Period: Overall Study
Arm/Group | TLT Treatment Group 1 (Active TLT Treatment) | TLT Treatment Group 2 (Placebo) | Pilot Study Treatment Group 1 | Pilot Study Treatment Group 2
Started | 10 | 11 | 4 | 3
Completed (1 active participant excluded as "completer" in analyses because last visit was out of window.) | 8 (1 completed study but was excluded as a "completer" from analyses because started a new treatment) | 8 (1 completed study but was excluded as a "completer" from analyses because started a new treatment) | 3 (1 non-completer included in analyses because only missed follow up, completed all treatment visits.) | 1 (Completer excluded from analyses because determined to be not eligible at end of study.)
Not Completed | 2 | 3 | 1 | 2
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0
Not completed — participant did not have time | 1 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: TLT: 3 randomized participants completed less than 4 treatments so they were not included in analyses. 9 participants screen failed. 5 participants decided not to participate after the screen (time commitment, no longer interested, etc). 1 participant was discontinued by the investigator pre-treatment - discovered that primary diagnosis was PTSD.
Groups:
- TLT Treatment Group 1: The TLT group will receive 2 near-infrared radiation via Transcranial LED Therapy (TLT) treatments per week for 8 weeks
  Near-infrared radiation via Transcranial LED Therapy: The subject will lie down comfortably on a exam bed . The sites of application of TLT (left and right forehead) will be inspected for any skin lesions (e.g. laceration or signs of inflammation) which would contraindicate the treatment. The subject will wear protective eyewear in the form of goggles or eye pads.
  The staff administering the TLT will be careful not to shine the light in or near the eyes of the subject. The two OLS devices will be secured in position with the use of a Hair Net. The delivery of the TLT is expected to last 20 min total (simultaneous application on the left and right forehead). The subject will be asked to rest for five minutes after the delivery of TLT. The skin at the sites of the application will be inspected again prior to dismissing the subject.
- Screen Fail/Not Randomized: 9 participants screen failed (3 had HAM-D scores that were below the threshold for study inclusion, 2 had bipolar disorder, 1 had active substance abuse, 1 had an exclusionary comorbid medical disorder, 1 did not pass drug screen, 1 was not depressed) . 5 participants decided not to participate after the screen (1 due to time commitment, 2 were no longer interested, 1 was moving away, and 1 was lost to follow up). 1 was discontinued by investigator pre randomization at Visit 1 because it was discovered at Visit 1 that the patient's primary diagnosis was PTSD (MDD was secondary). Additionally, the patient's trauma symptoms significantly interfered with their ability to complete the study tasks.
- Pilot Study Screen Fail/Not Randomized: 10 participants screen failed (5 had HAM-D scores that were above threshold for study inclusion criteria, 1 had too many failed trials in the current depressive episode, 1 had active substance abuse, 2 did not meet criteria for Major Depressive Disorder at the time of the screening visit, 1 had just started psychotherapy at the time of the screen). 1 participant dropped out pre-randomization due to time constraints.
  (see protocol change 10/28/2014)
- Total: Total of all reporting groups
Arm/Group | TLT Treatment Group 1 | TLT Treatment Group 2 | Screen Fail/Not Randomized | Pilot Study Treatment Group 1 | Pilot Study Treatment Group 2 | Pilot Study Screen Fail/Not Randomized | Total
Number analyzed (Participants) | 10 | 11 | 15 | 4 | 3 | 11 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 15 | 4 | 3 | 11 | 54
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12.8) | 50.7 (13.3) | 49.9 (10.8) | 47 (14) | 47.7 (13.5) | 38.3 (11.7) | 46.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 8 | 1 | 3 | 8 | 33
  Male | 4 | 4 | 7 | 3 | 0 | 3 | 21
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 15 | 4 | 3 | 11 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale (HAM-D 17) Score
Description: We anticipate that TLT will decrease HAM-D17 scores in study subjects significantly more than Sham treatment. We expect that we will be also able to estimate the effect size of the antidepressant action of TLT. Analyses were done for all evaluable subjects (participants who met the a priori cut-off of a minimum of 4 t-PBM sessions for inclusion in the study analyses) and treatment completers (participants followed for the entire 8-week study period and who received a clinical assessment immediately after).
  HAM-D17 questions are rated on a scale of 0-4 or 0-2 (total score: 0-50) with higher scores indicating more severe pathology. Scores typically fall into the following ranges: not depressed = 0-7; mildly depressed = 8-13; moderately depressed = 14-18; severely depressed = 19-22; very severely depressed = 23 and over.
  For the pilot study, we analyzed subjects from Baseline to Week 8. A last observation carried forward (LOCF) was performed to account for one week 8n missing value.
Time Frame: Visit 1 (Baseline) and Visit 17 (Week 9); Pilot Phase: Visit 1 (Baseline) and Week 8
Population: 3 randomized subjects excluded from TLT analyses because they received <4 t-PBM treatments. 2 study completers from Group 1(last visit out of window,started new treatment ),1 subject from Group 2(started therapy)excluded as completers in analyses. Pilot Study Treatment Group 2 excluded because there was no data(drop out, post screen ineligibility).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- TLT Treatment Group 1 (Active TLT Treatment) Completers: The TLT group will receive 2 near-infrared radiation via Transcranial LED Therapy (TLT) treatments per week for 8 weeks (completers only).
  Near-infrared radiation via Transcranial LED Therapy: The subject will lie down comfortably on a exam bed . The sites of application of TLT (left and right forehead) will be inspected for any skin lesions (e.g. laceration or signs of inflammation) which would contraindicate the treatment. The subject will wear protective eyewear in the form of goggles or eye pads.
  The staff administering the TLT will be careful not to shine the light in or near the eyes of the subject. The two OLS devices will be secured in position with the use of a Hair Net. The delivery of the TLT is expected to last 20 min total (simultaneous application on the left and right forehead). The subject will be asked to rest for five minutes after the delivery of TLT. The skin at the sites of the application will be inspected again prior to dismissing the subject.
- TLT Treatment Group 2 (Placebo) Completers: The sham group will receive 2 treatments of the sham device per week for 8 weeks. This only includes those who were followed for the entire 8-week study period and who received a clinical assessment immediately after.
  Sham device: The sham device does not emit near-infrared radiation.
- Pilot Study Treatment Group 1: The TLT group will receive 2 TLT treatments per week for 3 weeks followed by a cross-over phase (where no treatment is given), followed by 2 sham treatments per week for 3 weeks.
  1 participant was missing a final visit 8 value, so LOCF was used for this value.
  (see protocol change 10/28/2014)
Arm/Group | TLT Treatment Group 1 (Active TLT Treatment) | TLT Treatment Group 2 (Placebo) | TLT Treatment Group 1 (Active TLT Treatment) Completers | TLT Treatment Group 2 (Placebo) Completers | Pilot Study Treatment Group 1
Number analyzed (Participants) | 9 | 9 | 6 | 7 | 4
units on a scale | -11.7 (7.47) | -5.3 (7.03) | -15.7 (4.41) | -6.1 (7.86) | -6.75 (4.85)
Statistical Analysis 1: Comparison: TLT Treatment Group 1 (Active TLT Treatment) vs TLT Treatment Group 2 (Placebo); Test type: Superiority or Other; p = 0.04, t-test, 1 sided — a priori threshold for statistical significance: p≤0.05; We used a modified intent-to-treat approach with LOCF and unpaired Student's t-test (one-way), comparing the change in total severity score
Statistical Analysis 2: Comparison: TLT Treatment Group 1 (Active TLT Treatment) vs TLT Treatment Group 2 (Placebo); Test type: Superiority or Other; p = 0.08, t-test, 2 sided — a priori threshold for statistical significance: p≤0.05; Modified intent-to-treat approach with lost observation carried forward (LOCF) and a two-tailed t-test to compare the change in total severity score
Statistical Analysis 3: Comparison: TLT Treatment Group 1 (Active TLT Treatment) Completers vs TLT Treatment Group 2 (Placebo) Completers; This analysis includes only treatment completers (participants who who were followed for the entire 8-week study period and who received a clinical assessment immediately after); Test type: Superiority or Other; p = 0.01, t-test, 1 sided — a priori threshold for statistical significance: p≤0.05; One-tailed t-test to compare the change in total severity score for treatment completers
Statistical Analysis 4: Comparison: TLT Treatment Group 1 (Active TLT Treatment) Completers vs TLT Treatment Group 2 (Placebo) Completers; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.02, t-test, 2 sided — a priori threshold for statistical significance: p≤0.05; Two-tailed t-test to compare the change in total severity score for treatment completers
Statistical Analysis 5: Comparison: Pilot Study Treatment Group 1; By means of a paired t-test we tested the significance of the change in the mean HAM-D17 total score (from baseline) to week 8. Although the primary comparison was with the last assessment (week 8). A last observation carried forward (LOCF) was also performed to account for one missing value at week 8; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

2. Secondary Outcome: Systematic Assessment for Treatment Emergent Events-systematic Inquiry (SAFTEE-SI)
Description: To assess the safety and tolerability of TLT in depressed subjects: We predict that TLT will be safe and well-tolerated, as assessed by the SAFTEE-SI. We anticipate no significant differences between TLT and Sham in side-effects.The SAFTEE is a commonly used instrument developed by the NIMH and adapted into a self-report instrument. The version we used is the same used by the NIMH-sponsored CO-MED trial. It examines all possible treatment-emergent side effects and adverse symptoms, including suicidal thoughts and behaviors, and self-injurious behavior.
  The SAFTEE analyses are ongoing and will be reported in a second paper (they are not included in the primary outcomes paper). The single value analyzed is the total number of distinct treatment-emergent side-effects (a side effect is defined as any item on the SAFTEE for which severity increased by two or more levels from baseline to any visit) that occurred for each subject. Range: 0 to 165; higher values represent worse outcomes.
Time Frame: Assessed at odd-numbered Visits 1-17. The single value to be analyzed is the number of distinct side effects that occurred at least once during these assessment visits for each subject.
Population: 3 subjects excluded from TLT because they received <4 t-PBM treatments.1 excluded from Group 1 due to unreliable reporting.1 Group 1 and 1 Group 2 excluded due to no final visit score.1 excluded from Pilot Study Treatment Group 1 due to no final visit score.Pilot Study Treatment Group 2 excluded due to no data(drop out, post screen ineligibility).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TLT Treatment Group 1 (Active TLT Treatment) | TLT Treatment Group 2 (Placebo) | Pilot Study Treatment Group 1
Number analyzed (Participants) | 7 | 8 | 3
units on a scale | -17 (12.60) | -9.38 (20.33) | -10.33 (13.48)

3. Secondary Outcome: Number of Participants With Adverse Events
Description: To assess the safety and tolerability of the TLT in depressed subjects: We predict that the TLT will be safe and well-tolerated by depressed patients, as assessed by the following rating scales: ADVERSE EVENTS FORM. We anticipate no significant differences in between TLT and Sham treatment as concerns side-effects.
  Due to the small sample size and the variability of reported adverse events, we decided that descriptive reporting (i.e. reporting each subject's adverse events individually) was more appropriate than analysis. All adverse events were reported in the adverse events section. In the outcome measure data table below we report the number of participants in each group who experienced an adverse event.
Time Frame: Visits 1, 3, 5, 7, 9, 11, 13, 15, and 17
Population: 3 randomized subjects excluded from TLT analyses because they received <4 t-PBM treatments.
Measure: Count of Participants; unit: Participants
Arm/Group | TLT Treatment Group 1 | TLT Treatment Group 2 | Pilot Study Treatment Group 1 | Pilot Study Treatment Group 2
Number analyzed (Participants) | 9 | 9 | 4 | 3
Participants | 7 | 2 | 1 | 1

4. Post Hoc Outcome: Change in Quick Inventory of Depressive Symptomatology-Self Rated Scale (QIDS-SR) Score
Description: This is a brief (16-item) self-report inventory of core depressive symptoms such as sleep, depressed mood, appetite, concentration, suicidal ideation, interest, energy, psychomotor retardation or agitation. QIDS scores range from 0-27. Severity of depression can be judged based on the total score: 1-5 = No depression, 6-10 = Mild depression, 11-15 = Moderate depression. 16-20 = Severe depression, 21-27 = Very severe depression. Analyses were done for all evaluable subjects (participants who met the a priori cut-off of a minimum of four t-PBM sessions for inclusion in the study analyses) and treatment completers (participants who were followed for the entire 8-week study period and who received a clinical assessment immediately after). Pilot Study Group 2 excluded because no analyses were completed for this group (see participant flow)
Time Frame: Visit 1 (Baseline) and Visit 17 (Week 9)
Population: Excluded: 3 randomized subjects who had <4 t-PBM treatments; 1 from Group 1 (unreliable reporting); 2 from Group 1 (started new treatment),1 from Group 2 (started therapy). 1 from Pilot study group 1 (no final visit). Pilot Study Group 2 excluded because there was no data (2 subjects dropped out, 1 subject ineligible--see Participant Flow).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TLT Treatment Group 1 (Active TLT Treatment) | TLT Treatment Group 2 (Placebo) | TLT Treatment Group 1 (Active TLT Treatment) Completers | TLT Treatment Group 2 (Placebo) Completers | Pilot Study Treatment Group 1
Number analyzed (Participants) | 8 | 9 | 5 | 7 | 3
units on a scale | -5.9 (6.29) | -3.7 (2.91) | -9.8 (4.09) | -4.3 (3.04) | -2.33 (4.22)
Statistical Analysis 1: Comparison: TLT Treatment Group 1 (Active TLT Treatment) vs TLT Treatment Group 2 (Placebo); Test type: Superiority or Other; p = 0.18, t-test, 1 sided — a priori threshold for statistical significance: p≤0.05; Last observation carried forward (LOCF), one tailed t-test to compare change in QIDS score
Statistical Analysis 2: Comparison: TLT Treatment Group 1 (Active TLT Treatment) Completers vs TLT Treatment Group 2 (Placebo) Completers; This analysis includes only treatment completers (participants who who were followed for the entire 8-week study period and who received a clinical assessment immediately after). One treatment completer in Group 1 was excluded because they consistently skipped several answers across self-rated scales for the duration of the study; Test type: Superiority or Other; p = 0.01, t-test, 1 sided — a priori threshold for statistical significance: p≤0.05; One-tailed t-test to measure the change in QIDS score for treatment completers
Statistical Analysis 3: Comparison: TLT Treatment Group 1 (Active TLT Treatment) Completers vs TLT Treatment Group 2 (Placebo) Completers; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.02, t-test, 2 sided — a priori threshold for statistical significance: p≤0.05; Two-tailed t-test measuring change in QIDS score for treatment completers

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. Study clinicians inquired about any adverse events once a week for all 8 weeks of treatment. Clinicians also asked about adverse events at Visit 17 (follow up visit after the 8 week treatment).
Arm/Group | TLT Treatment Group 1 | TLT Treatment Group 2 | Pilot Study Treatment Group 1 | Pilot Study Treatment Group 2
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 7/10 | 2/11 | 1/4 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TLT Treatment Group 1 (N=10) | TLT Treatment Group 2 (N=11) | Pilot Study Treatment Group 1 (N=4) | Pilot Study Treatment Group 2 (N=3)
gastro-intestinal sickness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
restless sleep (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
headaches (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
taste illusion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
abdominal bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gout (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
self-harm (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
insomnia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
visual illusions (vivid colors) (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
decreased memory; word finding difficulties (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
left torso pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
belching (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pressure/pain on back of head during 4T Scan (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
dizziness/tingling sensation in head (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No